CLINICAL TRIAL: NCT03388112
Title: Effects of Probiotics on the Gut Microbiome of Infants Treated With Antibiotics
Brief Title: Shanghai Infants Gut Microbiome Associated Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Director, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHSYEK2017
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Gastrointestinal Microbiome
Keywords: Probiotics,Gut Microbiome,Antibiotics,Infants
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- antibiotics (No Intervention): the patients in this arm will not receive probiotics.
- probiotics concurrent with antibiotic (Experimental): the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis for 2 weeks concurrent with antibiotic.
  Interventions: Dietary Supplement: Probiotics
- probiotics after antibiotic (Experimental): the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis for 2 weeks after antibiotic.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis with does of 1.5*10^7CFU for 2 weeks
  Arms: probiotics after antibiotic; probiotics concurrent with antibiotic

SUMMARY:
The purpose of this study is to evaluate the effect of probiotics on the gut microbiome of infants treated with antibiotics.

DETAILED DESCRIPTION:
This study aims to examin the impact of probiotics under 2 separate conditions, probiotics concurrent administration with antibiotic and probiotics administration during the recovery phase.Birth,7 days,14 days(or 21 days) and 42 days data will be collected and put into analysis to provide somes suggestions on the probiotics use in the clinical for the infants treated with antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with infectious diseases treated with antibiotic

Exclusion Criteria:

* Gestational weeks <37
* Birth weight <2500g or ≥4000g
* History of asphyxia anoxia at birth
* With congenital metabolic diseases or hereditary diseases
* With gastrointestinal diseases

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
change from birth,7 days,14 days(or 21 days) on gut mcrobiome at 42 days | 42 days
  change of the gut mcrobiome will be calculated at 42 days in comparison with birth,7 days,14 days(or 21 days)

SECONDARY OUTCOMES:
change from birth on gut mcrobiome at 7 days | 7 days
  change of the gut mcrobiome will be calculated at 7 days in comparison with baseline
change from birth and 7 days on gut mcrobiome at 14 days(or 21 days) | 14 days（or 21days）
  change of the gut mcrobiome will be calculated at 14(or 21 days) in comparison with birth and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No